CLINICAL TRIAL: NCT07041489
Title: A Multi Center, Randomized, Double-Blind, Placebo-controlled Trial With Extension to an Open-Label Study to Evaluate the Safety and Efficacy of Xtressé™ Supplement + Serum Treatment Combination in Promoting Hair Growth in Women With Self-perceived Thinning Hair
Brief Title: Evaluating the Combined Use of Supplement and Serum in Promoting Hair Growth in Women With Self-perceived Thinning Hair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Clinical and Cosmetic Research (Other)
Collaborators: Restore Biologics Holdings, Inc. dba Xtressé (Industry); Xtressé (TM) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCCR 03-2025
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Hair Thinning
Keywords: hair thinning; thinning hair; hair loss; thin hair
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded in Part A followed by Open-label in Part B of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention Group - Part A and Part B (Active Comparator): 43 subjects will be randomized to this group and will receive Xtressé™ supplements + serum during the double-blinded Part A and open-label Part B of the study.
  Interventions: Dietary Supplement: Active Comparator- Xtressé™ Supplement and Serum
- Placebo Group- Part A (Placebo Comparator): 42 subjects will be randomized to this group and will receive Placebo supplements and serum in only Part A of the study.
  Interventions: Dietary Supplement: Placebo Comparator- Placebo Supplement and Serum
- Placebo Group- Part B (Active Comparator): 42 subjects will enter the open-labelled Part B of the study and will receive Xtressé™ supplements + serum.
  Interventions: Dietary Supplement: Active Comparator- Xtressé™ Supplement and Serum

INTERVENTIONS:
Dietary Supplement: Active Comparator- Xtressé™ Supplement and Serum — Participants will receive 3 month supplies 3 times during the study. Participants will apply serum and take supplements daily.
  Participants in the Intervention group will receive Xtressé™ Supplements and Serum in Part A and Part B of the study.
  Participants in the Placebo Group will receive Xtressé™ Supplement and Serum in Part B of the study only.
  Arms: Intervention Group - Part A and Part B; Placebo Group- Part B
Dietary Supplement: Placebo Comparator- Placebo Supplement and Serum — Participants will receive 3 month supplies 3 times during the study. Participants will apply serum and take supplements daily.
  Participants in the Placebo Group will receive Placebo Supplement and Serum in Part A of the study only.
  Arms: Placebo Group- Part A

SUMMARY:
The goal of this clinical trial is to test how safe and effective it is to improve hair growth using an active gummy and serum combination treatment when compared to an inactive treatment combination in women with self-perceived thinning hair.

The main questions this trial aims to answer are:

* to confirm using photograph analytics, how much hair growth has increased in a marked area when using active treatment versus inactive treatment, and
* participants assessment and satisfaction with the hair growth using scaled assessments.

Participants who qualify will be asked to complete 6 to 7 visits after voluntarily consent has been given. The study is divided into two parts. In Part A participants will be randomly given either active or inactive treatment to use over 3 months. After 3 months, all participants will enter Part B of the study and will be given active treatment to use over the final 6 months of the study.

DETAILED DESCRIPTION:
In the study, participants will be asked to complete the following:

* Provide basic personal information (including date of birth, gender, race and ethnicity)
* Provide their medical/ surgical history and perform a medical exam (including but not limited to symptom-directed physical exam, skin type, vital signs, height, weight, laboratory assessments and pregnancy test collection)
* Follow study rules such as avoiding certain medications and treatments
* Provide information on any medications, treatments or reactions that started after the study began
* Apply serum and take gummy treatment daily, including completing a treatment diary
* Allow clinical assessments and documentation of the treatment, such as photography, hair density measurements, any reactions or side effects

To qualify for this trial, participants must:

* be a female adult between 28 to 65 years of age
* have consistent self-perceived thinning hair.
* give voluntary written consent
* be willing to follow study instructions and complete study requirements, including maintaining current diet and hair care routine, not using non-approved lotions and creams on the treatments areas
* allow photographs of the front and top area of the scalp
* not be pregnant or breast feeding before and during the study and agree to use acceptable forms of birth control
* confirm they are not sensitive to any of the study treatment ingredients

A relatively small area will be shaved off-center and top of the scalp for a dot-tattoo placement and this marked area will be used for clinical assessments throughout the study.

All photographs of the treatment area collected during the study will be used as study data.

All participants have the right to refuse further participation in the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Female adults between 28-65 years of age with consistent self-perceived thinning hair.
* Ludwig Scale I or II (mild to moderate thinning hair loss), assessed clinically.
* Fitzpatrick Skin Types I to VI.
* Agree to maintain their current diet, medications, exercise routines, hair shampooing, and color treatment frequency for the duration of the study.
* Ability and willingness to comply with the study protocol including regular visits and product application.
* Written informed consent obtained, including written consent to allow photographs to be used as part of the study data and documentation.
* For females of childbearing potential, a negative pregnancy test at screening and commitment to effective contraception throughout the study (oral / implant/ injectable/ transdermal contraceptives, intrauterine device, condom, diaphragm, abstinence, or a monogamous relationship with a partner who has had a vasectomy) to avoid pregnancy-related hormonal changes affecting hair density.

Exclusion Criteria:

* Pregnant or lactating or planning to become pregnant.
* Changes in hormonal therapy within 6 months prior to enrollment and throughout the study.
* Use of other medical hair loss treatments (e.g., Minoxidil, Dutasteride, Finasteride, laser or light therapy) within 3 months prior to study start and throughout the study.
* Micro-needling, PRP, or any other physical treatment modality on the scalp (within 6 months prior to study start and throughout the study).
* Use of GLP-1 inhibitors (e.g., Semaglutide) within 6 months prior to study start and throughout the study.
* Known uncontrolled health conditions (e.g., thyroid disease, anemia) that could confound study outcomes.
* Known sensitivity to any of the ingredients in the study medication.
* In the investigator's opinion, evidence of unwillingness, or inability to follow the restrictions and requirements of the protocol and complete the study.
* Subject has any conditions, findings in history, physical exam or laboratory assessments, which in the opinion of the investigator, would exclude the subject from continuing in this study.
* Treatment with an experimental drug, biologic or device within 12 weeks of the screening visit.

Ages: 28 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 85 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Increase in hair density (hairs per cm²) measured as the within-subject change from baseline to Month 3, assessed via Canfield HairMetrix® phototrichogram analyses. | an average of 3 months
  Quantitative hair measurements calculated by analyzing the participants digital images.
Increase in hair density (hairs per cm²) Measured as the within-subject change from baseline to Month 9, assessed via Canfield HairMetrix® phototrichogram analyses. | Up to 9 months
  Quantitative hair measurements calculated by analyzing the participants digital images.
Participant self-assessment of hair growth and satisfaction, collected via validated questionnaires. | Up to 9 months
  Observations and changes noted in hair loss graded on a scale of 0 to 4, with 0 as none and 4 as a very severe outcome.
  Observations and changes noted in quality of life based on hair loss, outcomes graded between extremely affected and not at all.

SECONDARY OUTCOMES:
Increase in hair density as measured by SOCAi | Up to 9 months
  Changes to the appearance of hair will be captured using the SOCAi system.
Improvements in hair quality (e.g., thickness, strength) and volume, evaluated by blinded investigator assessments | Up to 9 months
  Observations and changes noted in hair quality graded on a scale of -3 to +3, with -3 as greatly worsened/ decreased, 0 as no change and +3 as significantly increased/ improved.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Leavitt, Study Director — Restore Biologics Holdings, Inc. dba Xtressé
Locations (2):
- United States (2):
  - Skin Wellness Dermatology, Birmingham, Alabama
  - Center for Clinical and Cosmetic Research, Aventura, Florida